CLINICAL TRIAL: NCT02715882
Title: Randomized Single-blind Placebo-controlled Clinical Study of Safety and Tolerability of CBLB502 as a Neo-adjuvant Treatment in Patients With Colorectal Cancer, With Different Doses and Regimens
Brief Title: Clinical Study of Safety and Tolerability of CBLB502 as a Neo-adjuvant Treatment in Patients With Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BioLab 612 LLC (Industry)
Collaborators: Cleveland BioLabs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BL612-CBLB502
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; TLR5; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — CBLB502

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 injection of CBLB502 0.35 μg/kg (Experimental): One subcutaneous injection of CBLB502 0.35 μg/kg (not more 30 μg/injection) or Placebo at Day 1 before tumor removal
  Interventions: Drug: CBLB502; Drug: Placebo
- 1 injection of CBLB502 0.45 μg/kg (Experimental): One subcutaneous injection of CBLB502 0.45 μg/kg (not more 40 μg /injection) or Placebo at Day 1 before tumor removal
  Interventions: Drug: CBLB502; Drug: Placebo
- 2 injections of CBLB502 0.35 μg/kg (Experimental): Two subcutaneous injections of CBLB502 0.35 μg/kg (not more 30 μg/injection) or Placebo at Day 1 and Day 4 before tumor removal
  Interventions: Drug: CBLB502; Drug: Placebo
- 2 injections of CBLB502 0.45 μg/kg (Experimental): Two subcutaneous injections of CBLB502 at 0.45 μg/kg (not more 40 μg /injection) or Placebo at Day 1 and Day 4 before tumor removal
  Interventions: Drug: CBLB502; Drug: Placebo

INTERVENTIONS:
Drug: CBLB502
  Other Names: Entolimod
Drug: Placebo
  Other Names: PBS; Phosphate buffer saline

SUMMARY:
Randomized Single-blind Placebo-controlled Clinical Study of Safety and Tolerability of CBLB502 as a Neo-adjuvant Treatment in Patients With Colorectal Cancer, With Different Doses and Regimens

ELIGIBILITY:
Inclusion Criteria:

1. Written Patient Informed Consent for participation in the study
2. Men and women in the age above 18 years
3. Patients with confirmed diagnosis of colorectal cancer, indication to scheduled surgery for primary tumor removal
4. Should not have any previous anticancer therapy
5. Patient's life expectancy more than 3 months
6. ECOG performance status 0-1
7. Adequate hepatic and renal function:

   * Total bilirubin ≤1.5 upper limit of normal (ULN)),
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN, regardless of the presence of liver metastases,
   * Creatinine ≤2 x ULN
8. Adequate cardiac function including:

   * LVEF ≥45 by echocardiogram (ECHO) or multi gated acquisition scan,
   * 12-lead electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention,
   * QTcB interval QT (QTc by Bazett's formula) < 470 msec and no history of Torsades des Pointes or other symptomatic QTcB abnormality,
   * Absence of orthostatic hypotonia
9. Negative testing for serological markers of HIV-infection, viral hepatitis В and С, syphilis
10. Content to use barrier contraception methods by male/female patient and his/her partner in the study period

Exclusion Criteria:

1. Inability to obtain written Informеd consent for participation in the study
2. History of cardiovascular abnormalities including any conditions stated below:

   * Myocardial infarction/stroke for the last 6 months,
   * Stable abnormalities in regional contractility,
   * Cardiac failure (NYHA functional class III-IV),
   * Confirmed cardiomyopathy,
   * Clinically significant arrhythmias including any conditions stated below:

     * QT prolongation syndrome,
     * History of II or III-degree AV-block,
     * Bradycardia (HR < 50 beats per min.) or tachycardia (HR >100 beats per min.)
   * Blood pressure abnormalities:

     * 2 degree uncontrolled arterial hypertension (systolic blood pressure > 160 mm Hg or diastolic blood pressure > 105 mm Hg),
     * Hypotension (systolic blood pressure < 90 mm Hg)
3. History of severe allergic, systemic and other oncologic diseases
4. Decompensated diabetes mellitus with glycolated hemoglobin level (HbA1c) > 7%
5. Administration of drug products with evident effect on immune system for previous 3 months prior screening (including corticosteroids. Remark: Topical agents (e.g. for rash treatment), inhalation aerosols (e.g. for treatment of broncho-obstructive diseases), eye drops and agents for local administration (e.g. to joint cavity) is allowed
6. Participation in other clinical studies or administration of study products for 30 days prior screening, or persisting adverse reactions of the study product
7. Patients that have not taken CBLB502
8. Patients with hypersensitivity/allergy to CBLB502 or excipients of the drug product; NSAID (including ibuprofen)
9. Pregnant or lactating women
10. History of salmonellosis
11. Body mass > 88 kg; no obesity which means BMI in the range 18.5-25 kg/m2 for women and 22-27 kg/m2 for men
12. Men and women of childbearing age which do agree to use double contraception method, oral contraception or abstain from sex contacts throughout the study
13. Alcohol abuse, drug abuse and any other medical, psychological and social reasons which may, in accordance with the investigator, affect patient's participation in the study, may prevent adequate assessment of the study results
14. Any conditions which are unstable or may endanger patient's safety and/or affect his/her adherence to the investigator instruction
15. Any patient is not able or willing to cooperate with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability evaluation as measured by adverse events and assessed as changes in vital signs and clinical laboratory measurements, physical examination findings and ECG readings | Baseline to up to 14 days after the drug administration

SECONDARY OUTCOMES:
Assessment of immune cells change in tumor by H&E and ICH staining | On Day 7 (Surgery day) after the drug administration
Determination of levels of cytokine IL-6 in blood by multiplex assays | Baseline to up to 7 days after the drug administration
Determination of levels of cytokine IL-8 in blood by multiplex assays | Baseline to up to 7 days after the drug administration
Determination of levels of cytokine IL-10 in blood by multiplex assays | Baseline to up to 7 days after the drug administration
Determination of levels of cytokine G-CSF in blood by multiplex assays | Baseline to up to 7 days after the drug administration
Determination of levels of cytokine TNFа in blood by multiplex assays | Baseline to up to 7 days after the drug administration
Specific T-cell responses measured by ELIspot | Baseline to up to 14 days after the drug administration
Antibody titer to CBLB502 as measured by ELISA | Baseline and on day 14 after the drug administration
Blood leukocytes by FACS | Baseline to up to 7 days after the drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Sergei I. Achkasov, MD PhD, Principal Investigator — Federal State Budgetary Institution "State Scientific Center of Coloproctology named after A.N. Ryzhikh" Ministry of Health of the Russian Federation; Nikolay V. Kislov, MD PhD, Principal Investigator — Federal State Institution of Health of the Yaroslav Region "Regional Clinical Oncology Hospital"; Sergei V. Odintcov, MD PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with polyclinic" Department of Presidential Affairs of the Russian Federation
Locations (1):
- Federal State Budgetary Institution "State Scientific Center of Coloproctology named after A.N. Ryzhikh" Ministry of Health of the Russian Federation, Moscow, Russia

REFERENCES:
- See also: Related Info — http://www.cbiolabs.com/cblb502